CLINICAL TRIAL: NCT06146582
Title: The Impact of a Personalized Care Intervention on 90-day Post-Discharge Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laguna Health, Inc (Industry)
Collaborators: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-003810
Record Dates: First submitted 2023-11-17; First posted 2023-11-24 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Cardiovascular Diseases
Keywords: Readmissions; Behavioral Health; Care Transitions; Social Determinants of Health; Contextualizing Healthcare; Virtual Coaching
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Participants were assigned upon consent randomly to an intervention or control group. The intervention group received support from Laguna Coaches and Laguna's mobile app for 90 days, the control group did not receive any support from Laguna coaches or Laguna's app.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Experimental): Group received support from Laguna Coaches
  Interventions: Behavioral: Laguna Coach and App Intervention Group
- Control Arm (No Intervention): Group received no support from Laguna Coaches

INTERVENTIONS:
Behavioral: Laguna Coach and App Intervention Group — Behavioral, mental and contextual support was delivered through personal interactions with Laguna Coaches via mobile app, phone, video, or web chat. Care interventions were individualized to best match each participant's needs and strengths. Support will be provided to participants through interactions over approximately 90 days.
  Arms: Intervention Arm

SUMMARY:
The purpose of this 90 day study is to demonstrate the extent to which participants with cardiovascular conditions can improve their recovery at home through a mobile app, support and resources made available to them after hospitalization. The study will evaluate the effectiveness of personal care intervention support, including one-on-one guidance, educational information, check-ins, and Laguna's mobile app to help participants recover better after hospitalization.

DETAILED DESCRIPTION:
This study was designed to provide support to a select group of participants by supplementing the hospital-provided discharge instructions. Laguna integrated hospital provided clinical guidance and Laguna's personalized contextual care protocols, with the goal of improving health outcomes and reducing readmissions within 90 days post-discharge.

Particiants in the intervention group received support from Laguna Health via Laguna's mobile app, phone, video, text, or web chat. Laguna provided contextual support to remove recovery barriers to these intervention participants.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to the hospital with a diagnosis of a cardiovascular disorder as defined by the coded diagnoses for that admission
* Discharged to home
* Converse in English
* Uses a telephone (landline or cell phone)

Exclusion Criteria:

* Participant unable to provide informed consent
* Participant lacks cognitive ability to participate in the study interventions as judged by the individual initiating the consenting process

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-12-29 (Actual)

PRIMARY OUTCOMES:
Unplanned All Cause Readmission Rate | 90 Days Post-Discharge

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P Olson, Ph.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD